CLINICAL TRIAL: NCT07301190
Title: First-in-Human Experience Using a Novel Shape-Adaptive Pulsed Field Ablation Catheter in Persistent Atrial Fibrillation
Brief Title: FIH Study of PFLotus in Persistent Atrial Fibrillation
Acronym: PFLotus- FIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Hanxiong Liu, Professor, The Third People's Hospital of Chengdu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFLotus- FIH
Record Dates: First submitted 2025-12-09; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; pulmonary vein isolation; ablation time; procedure time; freedom from atrial tachyarrhythmia recurrence; cavotricuspid isthmus ablation; mitral isthmus ablation; coronary sinus
MeSH Terms: conditions — Atrial Fibrillation | interventions — Irreversible Electroporation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation Group (Experimental): PVI was performed in all patients. Additional linear ablation strategies Including the left atrial posterior wall (LAPW), mitral isthmus (MI), or cavotricuspid isthmus (CTI), were performed at the operator's discretion.
  Interventions: Device: Pulse field ablation with the PFLotus catheter

INTERVENTIONS:
Device: Pulse field ablation with the PFLotus catheter — PVI was performed in all patients. Additional linear ablation strategies Including the left atrial posterior wall (LAPW), mitral isthmus (MI), or cavotricuspid isthmus (CTI), were performed at the operator's discretion.

SUMMARY:
Single-shot pulsed-field ablation (PFA) catheters maximize pulmonary vein isolation (PVI) efficiency but are limited for focal or linear ablation. The goal of this clinical trial is to evaluate the safety and effectiveness of a novel, PFA catheter that transitions between large 'petals' (single-shot), and a small, spherical 'bud' (large-focal/linear), enabling a PVI-plus strategy in patients with persistent AF (PersAF).

The main questions it aims to answer are:

1. Is there an absence of serious procedure or device-related adverse events within 7 days?
2. Can the catheter achieve durable lesions?

This trial enrolled patients with perAF , who were treated under general anesthesia with the shape-adaptive PFA catheter (PFLotus, bipolar, biphasic, 850 V, 60 μs, EnChannel Medical).

Participants will:

1. Undergo PVI and linear ablation with the PFLotus PFA catheter under general anesthesia;
2. Undergo remapping within 3-month post the index ablation to assess the durability of the lesions;
3. Undergo follow-up occurred at 7 days, 30 days, 3, 6, and 12 months. Recurrence was assessed via 12-lead ECG at each visit and 24-hour or 7-day Holter monitoring at 6 and 12 months.

DETAILED DESCRIPTION:
Background

Catheter ablation with thermal energy sources, including radiofrequency (RF) or cryoablation, is a well-established and effective treatment for atrial fibrillation (AF), demonstrating comparable safety and efficacy in studies where pulmonary vein isolation (PVI) is the procedural endpoint. However, the non-selective diffusion of thermal energy risks collateral damage to adjacent anatomical structures, a limitation for both clinical application and technological advancement. These two catheter types each present distinct trade-offs: point-by-point RF ablation requires considerable operator skill and longer procedure times, while cryoballoon ablation, though more user-friendly, lacks precise spatial control and is less suited for mapping and ablating non-PVI targets.

Pulsed field ablation (PFA) employs high-voltage, ultra-rapid electric fields to induce irreversible electroporation and cellular death. As a non-thermal modality, PFA demonstrates preferential selectivity for cardiomyocytes. This offers the potential to create durable lesions while better preserving surrounding critical structures such as the esophagus, blood vessels, pulmonary veins, and phrenic nerve. Notably, PFA has not been associated with thermal complications like atrioesophageal fistula, phrenic nerve palsy, or pulmonary vein stenosis, suggesting it may enhance PVI effectiveness while reducing procedural risks.

Current evidence for PFA in AF management stems largely from preclinical studies and single-arm clinical trials. Early first-in-human studies with various PFA systems have reported promising outcomes. In the pivotal single-arm PULSED AF trial, PFA (PulseSelect System, Medtronic) for paroxysmal and persistent AF yielded arrhythmia recurrence rates comparable to thermal ablation, with a low rate of primary safety events at one year. The MANIFEST-PF registry reported a 99.9% acute PVI success rate, very low major complications, and reduced atrial arrhythmia recurrence relative to thermal ablation.

A recent randomized controlled trial (RCT) in persistent AF (ADVENT trial) found PFA (Farapulse System, Boston Scientific) non-inferior to conventional thermal ablation for the primary efficacy endpoint-freedom from procedural failure and post-procedural atrial tachyarrhythmias. Another RCT in persistent AF (Sphere-Per-AF trial) confirmed that PFA (Sphere-9 System, Medtronic) was comparable to thermal ablation in both effectiveness and safety, with the added advantage of shorter procedure times.

New catheter designs continue to emerge. The multi-electrode, force-sensing PFA catheter (Globe, Kardium Inc.) was developed as a single-step PVI solution. More recently, a basket-balloon hybrid PFA catheter (Volt™, Abbott) has entered first-in-human trials, with preliminary data supporting its immediate efficacy and safety in persistent AF. A recent meta-analysis concluded that PFA is associated with shorter procedure times but longer fluoroscopy times, while showing no significant differences in complication rates or AF recurrence compared to thermal ablation.

Thus, this first-in-human study aims to evaluate the safety and effectiveness of a novel, PFA catheter that transitions between large 'petals' (single-shot), and a small, spherical 'bud' (large-focal/linear), enabling a PVI-plus strategy in patients with persistent AF (PersAF).

Methods Study Design This was a first-in-human, prospective, single-arm, single-center trial evaluating the safety and efficacy of a novel a novel shape-adaptive PFA ablation catheter in PersAF patients. The study was approved by the local Ethics Committee and conducted in accordance with the Declaration of Helsinki. All participants provided written informed consent.

Study Population Eligible patients were 18-75 years old with documented symptomatic PerAF (AF duration 7-365 days) who were refractory or intolerant to at least one Class I or III antiarrhythmic drug.

Procedural Workflow All procedures were performed under general anesthesia. The activated clotting time was maintained≥300 seconds. A decapolar catheter was positioned in the coronary sinus and a ventricular electrode in the right ventricle. Transseptal puncture was performed under fluoroscopic guidance.

An electroanatomic map of the left atrium and pulmonary veins was created using a PENTARAY® catheter and the CARTO 3 system (Biosense Webster). The PFA sheath was inserted and continuously flushed. The PFLutos catheter was advanced into the left atrium and navigated to target sites.

PVI was performed in all patients. Additional linear ablation strategies Including the left atrial posterior wall (LAPW), mitral isthmus (MI), or cavotricuspid isthmus (CTI), were performed at the operator's discretion. For MI ablation, if persistent epicardial connections were identified, adjunctive ablation within the coronary sinus was performed. After a 20-minute waiting period, isolation and block were reassessed.

Follow-up Post-ablation antiarrhythmic drug use was determined by the operator and typically discontinued after three months. Oral anticoagulation was maintained per guidelines. Structured follow-up occurred at 7 days and 3 months post-ablation, with lesion durability assessed via invasive remapping at 3 months. Additional visits were scheduled at 6 and 12 months. Atrial Tachyarrhythmia recurrence was assessed using 12-lead ECGs at each visit and 24-hour or 7-day Holter monitoring at 3, 6, and 12 months.

Endpoints The primary safety endpoint was the incidence of primary adverse events (PAEs) within 7 days post-ablation. Later-occurring events (device/procedure-related death, atrio-esophageal fistula, PV stenosis) were also classified as PAEs. Persistent diaphragmatic paralysis or phrenic nerve palsy at 3 months were considered PAEs.

The primary efficacy endpoint was acute procedural success, defined as the proportion of patients achieving: 1) complete electrical isolation of all PVs, and 2) for those undergoing linear ablation, confirmed bidirectional block at all targeted sites (LAPW, MI, CTI).

Secondary efficacy endpoints included:

1. Acute PV isolation success rate.
2. Acute success rate of bidirectional block for each linear ablation site.
3. Durable success rate of bidirectional block for each linear ablation site at 3-month remapping.
4. One-year freedom from atrial tachyarrhythmia recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years (inclusive), regardless of gender 2. Diagnosed with symptomatic persistent atrial fibrillation (AF). The patient's medical records document that the duration of AF episodes exceeds 7 days or the patient has a history of persistent AF, and meets **any one** of the following criteria:

1. A 24-hour ambulatory electrocardiogram (Holter) recorded within 365 days prior to enrollment shows AF throughout the monitoring period.
2. Two electrocardiograms (ECGs) obtained at an interval of more than 7 days within 365 days prior to enrollment both demonstrate AF.

3. Poor response to treatment with at least one class I or class III antiarrhythmic drug (AAD), or intolerance to class I or class III AADs.

4. Willing to participate in the trial, comply with the follow-up requirements specified in the protocol, and sign the informed consent form.

Exclusion Criteria:

1. Paroxysmal atrial fibrillation (AF)
2. AF caused by electrolyte disorders, thyroid diseases, or reversible/non-cardiac etiologies
3. Patients undergoing retreatment after ablation for rapid atrial tachyarrhythmias
4. Patients with sustained ventricular tachycardia or ventricular fibrillation
5. Left atrial anteroposterior diameter > 55 mm
6. Pulmonary vein (PV) stenosis (>70%) or prior PV stent implantation
7. History of left atrial ablation or cardiac surgery (including left atrial appendage closure)
8. Implantation of permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardioverter-defibrillator (with or without biventricular pacing function)
9. Contraindications to anticoagulation, or history of coagulation or bleeding abnormalities
10. Severe pulmonary disease: severe pulmonary arterial hypertension or any pulmonary disease with severe dyspnea involving blood gas abnormalities
11. Any of the following cardiac surgeries, implants, or conditions:

    * Prosthetic heart valve
    * NYHA Class III or IV congestive heart failure, or left ventricular ejection fraction (LVEF) < 40%
    * Atrial septal defect or ventricular septal defect closure
    * Atrial myxoma, left atrial appendage device implantation or occlusion
12. History of any of the following within 3 months prior to the procedure:

    * Myocardial infarction
    * Unstable angina
    * Percutaneous coronary intervention
    * Cardiac surgery (including coronary artery bypass grafting)
    * Hospitalization for heart failure
    * Pericarditis
13. History of any of the following within 3 months prior to the procedure:

    * Cerebral infarction or transient ischemic attack (TIA)
    * Documented thromboembolic events (e.g., confirmed by transesophageal echocardiography [TEE])
14. History of malignant tumor or expected life expectancy < 12 months
15. Mental disorders or history of mental illness with inability to cooperate independently
16. Lactating, pregnant, or women planning or potentially becoming pregnant
17. Acute or severe systemic infection, or significant abnormalities in liver/renal function
18. Participation in other interventional clinical trials, or ineligibility for enrollment as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint | Seven days post index ablation procedure
  The primary safety endpoint was the incidence of primary adverse events (PAEs) within 7 days post-ablation. Later-occurring events (device/procedure-related death, atrio-esophageal fistula, PV stenosis) were also classified as PAEs. Persistent diaphragmatic paralysis or phrenic nerve palsy at 3 months were considered PAEs.
The primary efficacy endpoint | Immediately after the index ablation procedure
  The primary efficacy endpoint was acute procedural success, defined as the proportion of patients achieving: 1) complete electrical isolation of all PVs, and 2) for those undergoing linear ablation, confirmed bidirectional block at all targeted sites (LAPW, MI, CTI).

SECONDARY OUTCOMES:
Rate of Acute Pulmonary Vein (PV) Isolation Success [Secondary Efficacy Endpoint] | Immediate after the index ablation procedure
  The outcome is defined as the proportion of participants who achieve complete electrical isolation of all targeted pulmonary veins immediately after the index ablation procedure.
Acute Bidirectional Block Success Rate for Each Targeted Linear Ablation Site [Secondary Efficacy Endpoint] | Immediate after the index ablation procedure
  The outcome is defined as the proportion of each targeted linear ablation site (e.g., left atrial posterior wall [LAPW], mitral isthmus [MI], cavotricuspid isthmus [CTI], superior vena cava [SVC]) that achieves verified bidirectional block immediately after the index ablation procedure. Each linear site is assessed independently, and the success rate for each site is reported separately.
Durable Bidirectional Block Success Rate for Each Targeted Linear Ablation Site at 3-Month Remapping [Secondary Efficacy Endpoint] | 3 months after the index ablation procedure
  The outcome is defined as the proportion of each targeted linear ablation site (LAPW, MI, CTI, SVC) that maintains verified bidirectional block (without recurrence of conduction) at 3-month remapping after the index ablation procedure. Each linear site is assessed independently, and the durable success rate for each site is reported separately.
1-Year Freedom from Atrial Tachyarrhythmia Recurrence [Secondary Efficacy Endpoint] | 1 year after the index ablation procedure
  The outcome is defined as the proportion of participants who remain free from recurrent atrial tachyarrhythmias (including atrial fibrillation, atrial flutter, atrial tachycardia) within 1 year after the index ablation procedure. Recurrence is defined as any episode of atrial tachyarrhythmia lasting ≥30 seconds, confirmed by 12-lead electrocardiogram or 72-hour Holter monitoring, following the 3-month blanking period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital of Chengdu, Chengdu, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD to be shared include baseline demographic and clinical data, procedural parameters (e.g., PFA settings, ablation sites), safety data (adverse events within 7 days and follow-up), effectiveness data, and post-PFA voltage mapping results. These IPD are all data used in the primary results publication, as sharing them supports reproducible research and advances the understanding the use of PFLotus PFA catheters in persistent AF.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2-year post primary publication
Access Criteria: 1. Eligible Recipients:
     Qualified researchers with academic/institutional affiliation, who submit a feasible research proposal and agree to comply with data protection regulations.
     Accessible MaterialsDe-identified individual participant data (baseline, procedural, follow-up data related to PFA/AF) and supporting documents (study protocol, statistical analysis plan, redacted clinical study report). Identifiable information and raw imaging data are excluded.
  2. Access Process Submit application (proposal, CV, IRB approval, signed DUA) to the corresponding author via designated email.